CLINICAL TRIAL: NCT05890547
Title: Recurrent Salivary Gland Infections in Covid-19
Acronym: RecSalivary
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Eslam Farid Abu Shady ,MD, lecturer, Benha University
Other Study IDs: RC 21-4-2023; Benha university (Other: Benha university)
Record Dates: First submitted 2023-06-02; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Recurrent Salivary Gland Infections in Covid-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Group (1) comprises 30 patients with Covid-19 infection representing the study group COVID-19 diagnosis will be based on a positive SARS-CoV-2 nasopharyngeal swab on real-time reverse transcription-polymerase chain reaction (RT-PCR) in the presence of clinical and/or radiological signs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: comprises 30 patients with Covid-19 infection representing the study group COVID-19 diagnosis will be based on a positive SARS-CoV-2 nasopharyngeal swab on real-time reverse transcription-polymerase chain reaction (RT-PCR) in the presence of clinical and/or radiological signs.
- Control group: comprises 30 patients without a history of Covid-19 infection as a control group.

SUMMARY:
The aim of this study is to find out the role of Covid-19 in salivary gland infection and its recurrence.

DETAILED DESCRIPTION:
This is a prospective clinical study of 60 patients. The study will be performed in the Otolaryngology department, Faculty of Medicine, Benha University during the duration from June 2023 to December 2023.

Inclusion criteria:

Adult patients aged ≥18 years.

Exclusion criteria:

* Patients with known autoimmune diseases,
* Diabetes Mellitus
* History of cancer in the region of the head and neck or previous radio and/or chemotherapy.
* History of facial nerve palsy,
* Oral and dental diseases including chronic sialadenitis or sialolithiasis.
* previous oral surgery.

Patients were divided into two equal groups each of 30 patients according to the cause of infection. Group (1) comprises 30 patients with Covid-19 infection representing the study group COVID-19 diagnosis will be based on a positive SARS-CoV-2 nasopharyngeal swab on real-time reverse transcription-polymerase chain reaction (RT-PCR) in the presence of clinical and/or radiological signs and group (2) comprises of 30 patients with non-Covid-19 infection as a control group.

All patients will be submitted to full ENT and intraoral clinical examination. We will Compare both groups as regards patients' characteristics, risk factors, etiology, symptoms, and rate of recurrence of sialadenitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years with a history of CIVID-19 infection in the study group and of similar age without a history of COVID-19 infection.

Exclusion Criteria:

* Patients with known autoimmune diseases,
* Diabetes Mellitus
* History of cancer in the region of the head and neck or previous radio and/or chemotherapy.
* History of facial nerve palsy,
* Oral and dental diseases including chronic sialadenitis or sialolithiasis.
* previous oral surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients aged ≥18 years with a history of CIVID-19 infection in the study group and of similar age without a history of COVID-19 infection.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
occurrence or recurrence of sialoadenitis | 6 months
  Compare both groups as regards patients' characteristics, risk factors, etiology, symptoms, and rate of recurrence of sialadenitis.

CONTACTS AND LOCATIONS:
Overall Officials: Eslam Abu Shady, MD, Principal Investigator — medical school
Locations (1):
- Benha university hospitals, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: Undecided